CLINICAL TRIAL: NCT05227365
Title: Treatment Evaluation of Neuromodulation for Tinnitus - Stage A3 (TENT-A3)
Brief Title: Treatment Evaluation of Neuromodulation for Tinnitus - Stage A3
Acronym: TENT-A3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Neuromod Devices Ltd. (Industry)
Collaborators: BRAI3N (clinical site), Belgium (Unknown); St. James's Hospital, Ireland (Other); German Hearing Center Hannover (clinical site), Germany (Unknown); Avania (CRO/project manager), Netherlands (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TENT-A3
Record Dates: First submitted 2022-01-26; First posted 2022-02-07 (Actual); Last update posted 2022-12-27 (Actual); Status verified 2022-12

CONDITIONS: Tinnitus
MeSH Terms: conditions — Tinnitus

STUDY DESIGN:
Intervention Model Description: Multi-site, single-arm repeated measures prospective investigation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Treatment Arm Study (Other): The Lenire device is a CE marked medical device intended to reduce the symptoms of tinnitus. It comprises a handheld controller, an intra-oral device called a Tonguetip that delivers gentle electrical stimulation to the tongue, and a set of wireless headphones that deliver audio stimulation to the ears. The sound and tongue stimulation are configured and calibrated to individual participant hearing and sensation characteristics during the initial fitting procedure completed by a trained clinician. The participants will receive 12 weeks of treatment, in which the first 6-weeks will consist of sound-only stimulation (PS6-No ETS) and the second 6-weeks will consist of bimodal stimulation (PS6, includes sound and tongue stimulation).
  Interventions: Device: Lenire

INTERVENTIONS:
Device: Lenire — The sound stimulus of PS6 is comprised of sequences of tones and is spectrally modified according to the participant's hearing thresholds so that different components of the sound stimulus can be sufficiently heard by the participant irrespective of their hearing characteristics (audiological profile). The tongue stimulus of PS6 is delivered by an array of electrical signals via 32 transmucosal electrodes contacting the anterodorsal surface of the tongue. The sound and tongue stimulus parameters are presented with certain stimulus rates and timing relationships between modalities.
  Other Names: Lenire treatment; Lenire device; Bimodal neuromodulation

SUMMARY:
TENT-A3 is a single arm repeated measures prospective investigation evaluating the safety and efficacy of the Lenire device for tinnitus treatment. The Lenire device provides non-invasive bimodal (sound and tongue) stimulation to alleviate the symptoms of chronic, subjective tinnitus. Participants presenting to one of the several study sites with a diagnosis of chronic subjective tinnitus who meet the inclusion criteria are enrolled in the investigation while the study site is active. The objective of TENT-A3 is to determine whether the addition of tongue stimulation to sound-only stimulation provides additional clinically significant improvements in tinnitus symptoms beyond that of the sound-only stimulation component of the bimodal treatment.

DETAILED DESCRIPTION:
Tinnitus is the perception of sound in the absence of a corresponding external acoustic stimulus. The condition is most commonly referred to as 'ringing in the ears' but symptoms can manifest as buzzing, hissing, clicking or other complex sounds. The condition affects approximately 10-15% of the global population. Many tinnitus sufferers report feeling distressed by their symptoms and report a resulting diminishment in their quality of life and that of their families. There are currently limited treatment options for those suffering from tinnitus. To address the unmet clinical need for a safe, effective, and scalable tinnitus treatment, Neuromod Devices developed a non-invasive bimodal (sound and tongue) stimulation device to alleviate the symptoms of chronic, subjective tinnitus. This CE marked device, known as Lenire, will be used in the TENT-A3 investigation, which is part of a series of bimodal neuromodulation investigations for the CE marked Lenire device for evaluating its safety and efficacy for tinnitus treatment. The Lenire device has three components: (1) headphones for presenting sound binaurally to the ears, (2) a tongue component for electrically stimulating the top surface of the tongue, and (3) a controller to control the stimulation patterns. TENT-A3 is a single arm repeated measures prospective investigation. Participants presenting to one of the several study sites with a diagnosis of chronic subjective tinnitus who meet the inclusion/exclusion criteria are enrolled in the investigation while the study site is active. The objective of TENT-A3 is to determine whether the addition of tongue stimulation to sound-only stimulation provides additional clinically significant improvements in tinnitus symptoms beyond that of the sound-only stimulation component of the bimodal treatment. Up to 112 participants are being enrolled in the study. Participants are involved with four visits that includes screening visit (up to 10 weeks before enrollment), enrollment visit (Week 0), interim visit (Week 6), and final visit (Week 12). Participants receive sound-only stimulation (PS6-No ETS: PS6 with No Electrical Tongue Stimulation) during Stage 1 (enrollment to interim vist) and bimodal stimulation (PS6) during Stage 2 (interim to final visit). Several outcome measures and evaluations are performed at each visit to assess the efficacy, safety, satisfaction, compliance and quality of life related to the Lenire treatment for tinnitus to address the primary, secondary and additional endpoints of the study.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and over at time of consent
* Ability to read and understand Dutch, Flemish, English or German (depending on the site)
* Willing and able to provide and understand informed consent
* Willing to commit to the full duration of the investigation
* Subjective tinnitus
* Tinnitus duration for greater than or equal to 3 months and less than or equal to 10 years at time of consent
* Baseline THI greater than or equal to 38

Exclusion Criteria:

* Subjective tinnitus, where pulsatility is the dominant feature (participant reported)
* Objective tinnitus, where the tinnitus is also observed by the examiner
* Commenced usage of hearing aid within the last 90 days
* Meniere's disease
* Hospitalization, or visit to a physician, for a head or neck injury, including whiplash, in the previous 12 months
* TMJ Disorder
* Pregnancy
* Oral piercings that cannot or will not be removed for the second stage of the investigation
* Neurological condition that may lead to seizures or loss of consciousness (e.g. epilepsy)
* Severe cognitive impairment based on MMSE (score less than 20)
* Participant with a pacemaker or other electro-active implanted device
* Abnormal findings following otoscopy/tympanometry that may be contributing to or causing the tinnitus as assessed by an Audiologist/ENT
* Initiated new prescription medications or medical treatments in the previous 3 months that may impact the outcomes of the investigation, by discretion of the investigator
* Ceased prescription medications or medical treatments in the previous 3 months that may impact the outcomes of the investigation, by discretion of the investigator
* STAI score of >120
* Current or previous involvement in medico-legal cases (self-reported)
* Participant previously diagnosed with psychosis or schizophrenia
* Participants diagnosed with burning mouth syndrome
* Previous use of Lenire
* Previous involvement in a clinical investigation for tinnitus or had an experimental/surgical treatment for tinnitus
* Hearing loss of greater than 80 dB HL in any test frequency in the set {2k,3k,4k,6k,8k} Hz or greater than 40 dB HL in the set {250,500,1k} Hz either unilaterally or bilaterally
* The site PI does not deem the candidate to be suitable for the investigation for other reasons not listed above

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2022-03-21 (Actual); Primary Completion 2022-09-06 (Actual); Study Completion 2022-10-25 (Actual)

PRIMARY OUTCOMES:
Tinnitus Handicap Inventory (THI) | Enrollment visit to final visit (Week 0 to Week 12)
  Responder rate in Stage 2 (the second 6-week period of treatment from interim visit to final visit comprising combined sound and tongue stimulation) compared to the point-estimate of the responder rate observed during Stage 1 (the first 6-week period of treatment from enrollment visit to interim visit comprising sound-only stimulation) based on THI.

SECONDARY OUTCOMES:
Tinnitus Functional Index (TFI) | Interim visit to final visit (Week 6 to Week 12)
  Changes in symptoms of tinnitus as measured by TFI from the interim visit to the final visit.

OTHER OUTCOMES:
Heath Utilities Index Mark III (HUI3) | Screening visit to final visit (Screening to Week 12)
  Changes in quality of life as measured by HUI3 from the screening visit to the interim visit and from the screening visit to the final visit.
Satisfaction Questions | Interim visit to final visit (Week 6 to Week 12)
  Participant satisfaction rates with treatment as measured by two satisfaction questions at the final visit.
Tinnitus severity analysis on primary outcome measure | Enrollment visit to final visit (Week 0 to Week 12)
  Primary outcome measure analyzed for different tinnitus severity groups based on clinically established THI categories (e.g., none/slight, mild, moderate, severe, catastrophic, THI >= 38, THI < 38)

CONTACTS AND LOCATIONS:
Overall Officials: Welmoed Gjaltema, Study Director — Avania, Netherlands; Michael Boedts, Principal Investigator — BRAI3N, Belgium; Guan Khoo, Principal Investigator — St. James's Hospital, Ireland; Thomas Lenarz, Principal Investigator — German Hearing Center Hannover, Germany
Locations (3):
- BRAI3N, Ghent, Belgium
- German Hearing Center, Hanover, Germany
- The Wellcome HRB Clinical Research Facility at St. James's Hospital, Dublin, Ireland

REFERENCES:
- [Background] Conlon B, Langguth B, Hamilton C, Hughes S, Meade E, Connor CO, Schecklmann M, Hall DA, Vanneste S, Leong SL, Subramaniam T, D'Arcy S, Lim HH. Bimodal neuromodulation combining sound and tongue stimulation reduces tinnitus symptoms in a large randomized clinical study. Sci Transl Med. 2020 Oct 7;12(564):eabb2830. doi: 10.1126/scitranslmed.abb2830. PMID 33028707